CLINICAL TRIAL: NCT04031768
Title: Rest Time Before Blood Pressure Measurement Trial
Brief Title: Best Rest: Rest Time Before Blood Pressure Measurement Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Vital Strategies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: IRB00214827
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Hypertension; Blood Pressure; Cardiovascular Diseases; Cardiovascular Risk Factor
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 0-2-5-5 minutes rest group (Other): The order of rest periods for participants randomized to this arm will be:
  0 minutes 2 minutes 5 minutes 5 minutes
  Interventions: Other: Timing of rest prior to blood pressure measurement
- 0-5-2-5 minutes rest group (Other): The order of rest periods for participants randomized to this arm will be:
  0 minutes 5 minutes 2 minutes 5 minutes
  Interventions: Other: Timing of rest prior to blood pressure measurement
- 2-0-5-5 minutes rest group (Other): The order of rest periods for participants randomized to this arm will be:
  2 minutes 0 minutes 5 minutes 5 minutes
  Interventions: Other: Timing of rest prior to blood pressure measurement
- 5-0-2-5 minutes rest group (Other): The order of rest periods for participants randomized to this arm will be:
  5 minutes 0 minutes 2 minutes 5 minutes
  Interventions: Other: Timing of rest prior to blood pressure measurement
- 2-5-0-5 minutes rest group (Other): The order of rest periods for participants randomized to this arm will be:
  2 minutes 5 minutes 0 minutes 5 minutes
  Interventions: Other: Timing of rest prior to blood pressure measurement
- 5-2-0-5 minutes rest group (Other): The order of rest periods for participants randomized to this arm will be:
  5 minutes 2 minutes 0 minutes 5 minutes
  Interventions: Other: Timing of rest prior to blood pressure measurement

INTERVENTIONS:
Other: Timing of rest prior to blood pressure measurement — Each participant will have 4 sets of 3 blood pressure measurements taken. The participants will be randomized to the order in which they rest prior to each set of measurements.

SUMMARY:
The objectives of this study are to:

1. Determine the impact of wait time before initiating BP measurement on BP variability
2. Determine the difference in BP variability between measurements by amount of initial rest.

The investigators also aim to:

1. To determine the total time required to obtain a BP measurement.

DETAILED DESCRIPTION:
Hypertension guidelines recommend a minimum of five minute rest time prior to blood pressure (BP) measurements obtained for screening, diagnosis and management of hypertension. This recommended wait time is often not adhered to and is cited as a barrier to regular screening due to length of time, clinic workflow and provider burden. It is unclear if BPs obtained at different rest intervals would provide clinically similar measurements. This study therefore aims to determine if BPs obtained immediately or after 2 minutes are rest are non-inferior to the BPs obtained after the guideline recommended 5 minutes of rest. It also aims to determine the time required to measure BP from start to finish, to allow for easier identification of other potential barriers to regular BP screening practices in busy clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years

Exclusion Criteria:

* Presence of the following on both arms: rashes, gauze dressings, casts, edema, paralysis, tubes, open sores or wounds, withered arms, A-V shunts, or if blood has been drawn from arm within last week.
* Being mentally impaired, pregnant.
* Arm circumference exceeding 50 cm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Difference in Systolic Blood Pressure (mmHg) | 90 minutes
  Comparison of the average of 3 systolic BP measurements (mmHg) measured after 5 minutes rest with the average of 3 systolic blood pressure (SBP) measured after the other periods of rest (0 minutes, 2 minutes, second 5 minutes of rest)
Difference in Diastolic Blood Pressure (mmHg) | 90 minutes
  Comparison of the average of 3 diastolic BP measurements (mmHg) measured after 5 minutes rest with the average of 3 diastolic blood pressure (DBP) measured after the other periods of rest (0 minutes, 2 minutes, second 5 minutes of rest)

SECONDARY OUTCOMES:
Blood Pressure Variability (mmHg) | 90 minutes
  Difference between individual systolic and diastolic BP measurements (BP reading 1 - BP reading 2; BP reading 2 - BP reading 3) obtained per each rest period
Standard Deviation of Blood Pressures (mmHg) | 90 minutes
  Difference in standard deviation of the mean of 3 systolic and diastolic BPs obtained at each rest period
Coefficient of Variation of Blood Pressures | 90 minutes
  Difference in coefficient of variation (SD/mean) of 3 systolic and diastolic BPs obtained at each rest period

OTHER OUTCOMES:
Total time required to obtain a BP measurement (seconds) | 90 minutes
  For each rest time assignment, mean time from:
  * Seating -> cuff placement
  * Cuff placement -> first measurement
  * Start of cuff inflation to measurement completion/BP output on device
  * Overall: Time from seating -> completion of all 3 BP measurements, 30 seconds apart.

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Brady, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine Division of Pediatric Nephrology, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brady TM, Charleston J, Ishigami J, Miller ER 3rd, Matsushita K, Appel LJ. Effects of Different Rest Period Durations Prior to Blood Pressure Measurement: The Best Rest Trial. Hypertension. 2021 Nov;78(5):1511-1519. doi: 10.1161/HYPERTENSIONAHA.121.17496. Epub 2021 Oct 4. PMID 34601959